CLINICAL TRIAL: NCT02827175
Title: Evaluation of the Effectiveness of a Diagnostic Kit in the Etiological Diagnosis of Fevers of the Traveler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-45; 2013-A01536-39 (Other: idrcb)
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Fevers of the Traveler
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fevers of the travelers (Experimental)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Annually about 10 to 15 million international travelers from Europe visit tropical countries. Returning from a journey, fever is the cardinal symptom of many infections. This is the second reason for consultation (23%) for return from a trip, after digestive disorders (42%). Urgent evaluation must always be proposed. Although that may be the manifestation of a benign disease, fever of return can also presage a rapidly progressive and lethal disease. In 50% of cases, patients return home, after treatment and disappearance of symptoms, though the microorganism responsible for the pathology is not able to be identified. The prescription of a series of systematic biological examinations in the form of a diagnostic kit has shown its relevance and its effectiveness in improving the etiological diagnosis of endocarditis and pericardites for optimal support. In this study we propose to assess the effectiveness of the systematic prescription of a diagnostic kit 'fever of the traveler' to all patients hospitalized with a fever after returning from a trip. "Ready to use" kit brings together in a single bag (i) instructions for use, (ii) the tubes, bottles and jars for the etiological diagnosis of fever of the traveler in the usual support (iii) an additional blood tube for research of pathogens emerging.

Primary:

To assess the effectiveness of a diagnostic kit for the etiological diagnosis of fevers of travelers on the return.

Hypothesis:

Improvement of at least 15% of the etiological diagnosis of fevers of travelers on the return through the development of a diagnostic kit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a T >38.5 ° C with or without associated clinical signs.
* Patient who traveled outside metropolitan France within 45 days with the hospitalization.
* Patient is more than 18 years old.
* Patient who accept to have his medical records reviewed for research.
* Patient with health insurance

Exclusion Criteria:

* a feverish syndrome beyond 45 days after the return of their journey.
* a clinical symptomatologie on the return to journey without associated fever,
* minor(miner) ( 18 years).
* Pregnant or breast-feeding woman.
* Incapable major patient or outside state to express its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Number of etiological diagnosis established in relation to the number of prescribed kits | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Asssitance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided